CLINICAL TRIAL: NCT00633672
Title: A Comparative Efficacy and Safety Study of Nexium Delayed-Release Capsules (40mg qd and 20mg qd) Versus Ranitidine 150mg Bid for the Healing of NSAID-Associated Gastric Ulcers When Daily NSAID Use is Continued
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SH-NEN-0006
Record Dates: First submitted 2008-02-27; First posted 2008-03-12 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: NSAID Associated Gastric Ulcers
Keywords: NSAID; Nexium; esomeprazole; Gastric Ulcers
MeSH Terms: conditions — Stomach Ulcer | interventions — Esomeprazole; Ranitidine

ARMS (3):
- 1 (Experimental): 20mg Oral tablet daily
  Interventions: Drug: Esomeprazole
- 2 (Experimental): 40mg oral tablet daily
  Interventions: Drug: Esomeprazole
- 3 (Active Comparator): 150mg oral twice daily
  Interventions: Drug: Ranitidine

INTERVENTIONS:
Drug: Esomeprazole — 20mg Oral tablet once daily
  Other Names: Nexium
  Arms: 1
Drug: Ranitidine — 150mg oral twice daily
  Other Names: Zantac
  Arms: 3
Drug: Esomeprazole — 40mg oral tablet once daily
  Other Names: Nexium
  Arms: 2

SUMMARY:
Nonsteroidal anti-inflammatory drugs (NSAIDS) are often associated with gastric ulcers. This study looks at the treatment of these gastric ulcers with one of the three following treatment groups: esomeprazole 40 mg once daily; esomeprazole 20 mg once daily; or ranitidine 150 mg twice daily.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of a chronic condition (eg osteoarthritis or rheumatoid arthritis) that requires daily NSAID treatment for at least 2 months.
2. Other key inclusion criteria, as specified in the protocol.

Exclusion Criteria:

1. History of esophageal, gastric or duodenal surgery, except for simple closure of an ulcer.
2. History of severe liver disease, including (but not limited to) cirrhosis and acute or chronic hepatitis.
3. Other conditions and criteria, as specified in the protocol.

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2001-02; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
To assess the safety and efficacy of esomeprazole 40 mg qd versus ranitidine 150 mg bid through 8 weeks of treatment for the healing of gastric ulcers in patients receiving daily NSAID therapy. Healing is defined as the absence of gastric ulcers.

SECONDARY OUTCOMES:
Patient and investigator assessed GI symptoms for up to 8 weeks of treatment. | Assessments at week 0, week 4 and week 8
Safety and tolerability of the treatments for 8 weeks of treatment. | Assessments at week 0, week 4 and week 8

CONTACTS AND LOCATIONS:
Overall Officials: Paula Fernstrom, Study Director — Nexium Global Product Director, AstraZeneca